CLINICAL TRIAL: NCT06555510
Title: Preoperative Edema is a Significant Risk Factor for Post-hepatectomy Complications Regardless of the Underlying Disease.
Brief Title: Preoperative Edema is a Significant Risk Factor for Post-hepatectomy Complications
Status: Completed | Type: Observational
Sponsor: Kochi University (Other)
Responsible Party: Principal Investigator, Takehiro Okabayashi, Head of Gastroenterological Surgery, Kochi University
Other Study IDs: KHSC2401
Record Dates: First submitted 2024-08-06; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Patients Who Underwent Hepatectomy for Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: InBody — Bioelectrical impedance analysis

SUMMARY:
Aims: The relationship between bioelectrical impedance analysis (BIA) results and post-hepatectomy complications is unknown. This study aimed to identify the risk factors for post-hepatectomy complications from the BIA results.

Methods: This prospective, observational cohort study reviewed the data of patients who underwent hepatectomy between March 2018 and December 2022. The patients were matched using the following propensity score covariates: biliary enteric anastomosis and major hepatectomy. Risk factors for postoperative complications were investigated in a matched cohort.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of liver neoplasms

Exclusion Criteria:

* a body weight loss of >10% during the 6 months before surgery; the presence of distant metastases; or seriously impaired function of vital organs because of respiratory, renal, or heart disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We prospectively reviewed consecutive patients who underwent hepatectomy at the Kochi Health Sciences Center. Patients who underwent hepatectomy, regardless of the underlying disease, between March 2018 and December 2022 were eligible for the study. Patients who did not undergo preoperative BIA were excluded. Those who underwent repeat hepatectomies were included; however, if they underwent more than two hepatectomies in the study period, only the clinical features during the first hepatectomy period were included and those during the second or third hepatectomy period were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 414 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
incidence of post-hepatectomy complications | incidence of post-hepatectomy complications
  through study completion, 1year

CONTACTS AND LOCATIONS:
Locations (1):
- Takehiro Okabayashi, Kochi, Japan